CLINICAL TRIAL: NCT05515328
Title: Investigation of Metabolism and Pharmacokinetics and Absolute Bioavailability of BI 685509 (C-14) After Intravenous and Oral Administration in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How BI 685509 is Processed in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1366-0008; 2022-001549-19 (EudraCT Number)
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: The study has two parts:
  Part A: open-label, single-arm, single dose trial, Part B: non-randomised, open-label, fixed sequence crossover trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A: Arm 1 (Experimental)
  Interventions: Drug: [¹⁴C] BI 685509 formulation 1
- Part B: Arm 1 - Reference (Experimental)
  Interventions: Drug: [¹⁴C] BI 685509 formulation 2
- Part B: Arm 2 - Treatment (Experimental)
  Interventions: Drug: BI 685509 formulation 3

INTERVENTIONS:
Drug: [¹⁴C] BI 685509 formulation 1 — [¹⁴C] BI 685509 formulation 1
  Arms: Part A: Arm 1
Drug: [¹⁴C] BI 685509 formulation 2 — [¹⁴C] BI 685509 formulation 2
  Arms: Part B: Arm 1 - Reference
Drug: BI 685509 formulation 3 — BI 685509 formulation 3
  Arms: Part B: Arm 2 - Treatment

SUMMARY:
The main objective of Part A is to investigate basic pharmacokinetics of BI 685509 and total radioactivity, including mass balance, excretion pathways and metabolism following administration of BI 685509 to healthy male subjects.

The main objective of Part B is to determine the absolute bioavailability of BI 685509 after administration to healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP)), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 weight divided by height squared (kg/m2) (inclusive)
* Signed and dated written informed consent in accordance with International Council on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Male subjects with women of child-bearing potential (WOCBP) partner who are vasectomised or willing to use male contraception (condom or sexual abstinence) from time point of study drug administration until 15 weeks thereafter

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 40 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
Part A: fraction of [¹⁴C] radioactivity excreted into urine given as percentage of the administered dose in the time interval from 0 to last quantifiable time point (fe urine,0-tz) | up to 14 days
Part A: fraction of [¹⁴C] radioactivity excreted into feces given as percentage of the administered dose in the time interval from 0 to last quantifiable time point (fe feces,0-tz) | up to 14 days
Part B: Absolute bioavailability of BI 685509 (%, obtained from a ratio of dose normalised values of AUCo-∞ after [¹⁴C] BI 685509 formulation 2 and BI 685509 formulation 3 administration) | up to 4 days
  AUCo-∞: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity

SECONDARY OUTCOMES:
Part A: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC₀-tz) | up to 14 days
Part A: Maximum measured concentration of the analyte in plasma (Cₘₐₓ) | up to 14 days
Part B: Area under the concentration-time curve of [¹⁴C] BI 685509 formulation 2 and BI 685509 formulation 3 in plasma over the time interval from 0 to the last quantifiable time point (AUC₀-tz) | up to 4 days
Part B: Area under the concentration-time curve of [¹⁴C] BI 685509 formulation 2 and BI 685509 formulation 3 in plasma over the time interval from 0 extrapolated to infinity (AUC₀-∞) | up to 4 days
Part B: Maximum measured concentration of [¹⁴C] BI 685509 formulation 2 and BI 685509 formulation 3 in plasma (Cₘₐₓ) | up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Joseph D, Wong D, Mitra P, Auclair AM, Wolfgang T, Gao E, Herich L, Tiessen R. Mass balance and absolute bioavailability of avenciguat (14C) after intravenous or oral administration in healthy male participants. Expert Opin Investig Drugs. 2026 Jan 13:1-10. doi: 10.1080/13543784.2025.2612329. Online ahead of print. PMID 41489441
- See also: Related Info — http://www.mystudywindow.com